CLINICAL TRIAL: NCT04322526
Title: Naltrexone-induced Blockade of Neural Responses Induced by Fast-Acting Antidepressant Effects
Brief Title: Study of Naltrexone-Induced Blockade of Antidepressant Effects
Acronym: SONRISA2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marta Peciña, MD PhD (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Marta Peciña, MD PhD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO16050133
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Naltrexone; Tablets

STUDY DESIGN:
Intervention Model Description: This is a pharmaco-fMRI study of one single dose of naltrexone or placebo followed by an fMRI session in a crossover design.
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naltrexone, then placebo (Experimental): Naltrexone is thought to strongly block μ-opioid receptors. Oral (pill) opioid antagonist which will be used to modulate neural responses during the Contextual Framing and the Antidepressant fMRI Task.
  Interventions: Drug: Naltrexone 50 Mg Oral Tablet; Drug: Placebo oral tablet
- Placebo, then naltrexone (Placebo Comparator): In the naltrexone condition, participants will receive one tablet of 50mg Naltrexone hydrochloride.
  Interventions: Drug: Naltrexone 50 Mg Oral Tablet; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Naltrexone 50 Mg Oral Tablet — Naltrexone hydrochloride (ReVia®. Toronto, ON: Teva Canada Limited; 2015) (onset of action: ≥15 minutes; peak effect: ~1 hour; duration: ~24 hours).
Drug: Placebo oral tablet — Placebo tablet that has no inherent power to produce an effect. In the inert pill condition, participants will receive an oral placebo tablet.

SUMMARY:
The goal of this study is to determine whether antidepressant placebo effects and contextual cues broadly, can be blocked by one single dose of the µ-opioid antagonist naltrexone. To test this hypothesis, un-medicated, patients with MDD completed a randomized, double-blind, placebo-controlled, cross-over study of 50mg of the µ-opioid antagonist naltrexone or matching placebo, immediately before a Pharmaco-fMRI scanning session.

DETAILED DESCRIPTION:
Neuroimaging offers a precise and objective way to characterize the neural and molecular basis of the antidepressant response in humans. Furthermore, the combination of neuroimaging with pharmacological manipulations opens the possibility of investigating drug-induced brain changes associated with behavioral responses.

In this study, the investigators aimed to whether antidepressant placebo effects and contextual cues broadly can be blocked by one single dose of the µ-opioid antagonist naltrexone. To assess trial by trial manipulation of antidepressant placebo effects inside of the scanner, the investigators have developed and piloted an fMRI task, specifically designed to record and modulate mood improvement using simulated neurofeedback. In a pilot study using this task, patients with MDD who reported acute mood improvement in response to positive neurofeedback, showed increased blood-oxygen-level-dependent (BOLD) responses in the ACC, and in particular, the rostral ACC (rACC), a reliable marker of treatment response in depression, and analgesic effects. In summary, these preliminary studies demonstrate 1) the contribution of the opioid system to the formation of antidepressant effects in MDD; and 2) increased rACC BOLD responses in patients who reported acute mood improvement induced by positive neurofeedback after a fast-acting antidepressant.

Still, the opioid modulation of acute mood improvement and rACC BOLD responses in patients with MDD has not been investigated, which justifies the research proposed in this application. Based on this preliminary evidence, The investigators hypothesize that antidepressant effects in patients with Major Depression rely on opioid modulation of rACC activity, and therefore can be partially or totally blocked using the selective µ-opioid antagonist naltrexone.To test this hypothesis, 20 un-medicated, patients with MDD completed a randomized, double-blind, placebo-controlled, cross-over study of 50mg of the µ-opioid antagonist naltrexone or matching placebo, immediately before a Pharmaco-fMRI scanning session. The study aims to:

AIM 1: Evaluate the effect of naltrexone on acute mood improvement and rostral anterior cingulate (rACC) BOLD activity induced by positive neurofeedback after a fast-acting antidepressant. The investigators hypothesize that naltrexone-induced blockade of µ-opioid receptors will reverse the acute mood improvement and increased rACC BOLD activity induced by positive neurofeedback.

AIM 2: Determine the extent to which individual differences in the rACC BOLD activity induced by positive neurofeedback after a fast-acting antidepressant predict acute mood improvement. The investigators hypothesize that increased rACC BOLD activity induced by positive neurofeedback will be associated with greater acute mood improvement.

AIM 3: Define the role of the rACC BOLD activity induced by positive neurofeedback as a mediator of the effect of group (naltrexone versus placebo) in acute mood improvement.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18-55 years; fluent in English and with the capacity to understand the nature of the study and sign the written informed consent since the research instruments used in this study are not available in other languages;
* Written informed consent obtained;
* Outpatients with a current primary diagnosis of nonpsychotic Major Depressive Disorder (MDD) per the Mini-International Neuropsychiatric Interview (M.I.N.I) with or without certain anxiety disorders (e.g., generalized anxiety, panic, agoraphobia, social phobia, and specific phobia); HDRS-17 score of ≥ 16 at Screening Visit;
* No more than one failed antidepressant trial of adequate dose and duration, as defined by the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH-ATRQ);
* Participants will need to be antidepressant medication-free for at least 21 days prior to the collection of imaging data (five weeks for fluoxetine). However, individuals currently taking antidepressants will not be eligible to enroll in the study, even if they are willing to stop their medications.

Exclusion Criteria:

* Currently taking opioid analgesics or in acute opioid withdraw.
* Pregnant or breastfeeding or plan to become pregnant over the duration of the study;
* History (lifetime) of psychotic depressive, schizophrenic, bipolar (I, II, or NOS), schizoaffective, or other Axis I psychotic disorders;
* Meeting M.I.N.I. criteria for substance dependence in the last 6 months, except for nicotine, or substance abuse in the last 2 months;
* Requiring immediate hospitalization for psychiatric disorder or have an unstable general medical condition (GMC) that will likely require hospitalization or to be deemed terminal (life expectancy < 6 months after study entry);
* Requiring medications for their GMCs that contraindicate treatment with naltrexone;
* Having epilepsy or other conditions requiring an anticonvulsant;
* Receiving or have received during the current episode vagus nerve stimulation, ECT, or rTMS.
* Currently taking any psychiatric medication or other potential augmenting agents (e.g., T3 in the absence of thyroid disease, lithium, buspirone); Taking thyroid medication for hypothyroidism may be included only if they have been stable on the thyroid medication for 3 months;
* Receiving therapy that is depression specific, such as CBT or Interpersonal Psychotherapy of Depression (participants can participate if they are receiving psychotherapy that is not targeting the symptoms of depression, such as supportive therapy, marital therapy);
* Currently actively suicidal or considered a high suicide risk;
* Currently enrolled in another study, and participation in that study contraindicates participation in this study;
* Any reason not listed herein yet, determined by the site PI and research staff that makes participation in the study hazardous.
* Having any contraindication for the performance of an MRI, such as: the presence of metal implants or foreign metallic objects (e.g., braces or extensive dental work), severe claustrophobia, or inability to tolerate the scanning procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Peciña, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Bellefield Towers, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NIfTI-formatted images for imaging, documentation, and code (https://github.com/) developed as part of this project will be shared upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately following publication upon request. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Derived] Chen J, Mizuno A, Lyew T, Karim HT, Karp JF, Dombrovski AY, Pecina M. Naltrexone modulates contextual processing in depression. Neuropsychopharmacology. 2020 Nov;45(12):2070-2078. doi: 10.1038/s41386-020-00809-2. Epub 2020 Aug 25. PMID 32843703

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone, Then Placebo: In the naltrexone and then placebo arm, participants receive one-dose naltrexone 50mg one hour before a first fMRI scanning session on visit 1 followed by a one-dose placebo pill one hour before a second fMRI scanning session on visit 2.
  Naltrexone 50 Mg Oral Tablet: Naltrexone hydrochloride (ReVia®. Toronto, ON: Teva Canada Limited; 2015) (onset of action: ≥15 minutes; peak effect: ~1 hour; duration: ~24 hours).
  Placebo oral tablet: Placebo tablet that has no inherent power to produce an effect. In the inert pill condition, participants will receive an oral placebo tablet.
- Placebo, Then Naltrexone: In the placebo and then naltrexone arm, participants receive one-dose of placebo pill one hour before a first fMRI scanning session on visit 1 followed by a one-dose naltrexone 50mg one hour before a second fMRI scanning session on visit 2.
  Naltrexone 50 Mg Oral Tablet: Naltrexone hydrochloride (ReVia®. Toronto, ON: Teva Canada Limited; 2015) (onset of action: ≥15 minutes; peak effect: ~1 hour; duration: ~24 hours).
  Placebo oral tablet: Placebo tablet that has no inherent power to produce an effect. In the inert pill condition, participants will receive an oral placebo tablet.
Period: First Intervention (1 Day)
Arm/Group | Naltrexone, Then Placebo | Placebo, Then Naltrexone
Started | 13 | 12
Completed | 12 | 11
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Washout (1 Week)
Arm/Group | Naltrexone, Then Placebo | Placebo, Then Naltrexone
Started | 12 | 11
Completed | 11 | 9
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Period: Second Intervention (1day)
Arm/Group | Naltrexone, Then Placebo | Placebo, Then Naltrexone
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone, Then Placebo | Placebo, Then Naltrexone | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (5.2) | 25.9 (8.2) | 25.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: BOLD Responses in the rACC Cortex During the Processing of Contextual Cues at Baseline (Post-placebo)
Description: In order to identify the neural correlates of contextual processing, we examined changes in blood oxygenation level-dependent (BOLD) signal during the post-placebo fMRI scanning session.
Time Frame: [Approximately at day 1, 7]
Population: The goal of aim one was to identify the neural correlates of antidepressant placebo effects. This aim was accomplished by examining the neural responses to the Antidepressant placebo fMRI task during the placebo session only, regardless of whether participants were assigned to the placebo-naltrexone or the naltrexone-placebo intervention.
Measure: Mean (Standard Deviation); unit: BOLD signal
Groups:
- fMRI BOLD Responses in the rACC Cortex (Placebo Session): We examined baseline brain measures of contextual processing during the placebo session only. In particular, we obtained whole-brain BOLD fMRI responses during the processing of contextual cues and extracted BOLD signal measures in the rACC.
  Post-naltrexone brain responses were not used for this analysis.
Arm/Group | fMRI BOLD Responses in the rACC Cortex (Placebo Session)
Number analyzed (Participants) | 20
BOLD signal | 0.47 (0.76)
Statistical Analysis 1: Comparison: fMRI BOLD Responses in the rACC Cortex (Placebo Session); Changes in BOLD signal in the rACC during the processing of contextual cues (pleasant > unpleasant); Test type: Other; p = 0.01, t-test, 2 sided

2. Primary Outcome: Naltrexone-induced Changes in BOLD Responses in the rACC Cortex During the Processing of Contextual Cues (Placebo vs. Naltrexone)
Description: In order to identify naltrexone-induced changes in the neural correlates of contextual processing, we examined changes in blood oxygenation level-dependent (BOLD) during the fMRI scanning session between Naltrexone vs. placebo pill.
Time Frame: [Approximately at day 1, 7]
Population: The goal of aim two was to investigate the effects of one single dose of naltrexone on the neural correlates of antidepressant placebo effects. This aim was accomplished by examining changes in the neural responses to the Antidepressant placebo fMRI task from the naltrexone to the placebo session, regardless of the order of each intervention.
Measure: Mean (Standard Deviation); unit: changes in BOLD signal
Groups:
- fMRI BOLD Responses in the rACC Cortex (Naltrexone vs Placebo): We examined naltrexone-induced changes in brain signal during the processing of contextual cues by extracting brain responses in the rACC and comparing then during the baseline (placebo only) and the naltrexone session using paired-t test statistical analysis.
Arm/Group | fMRI BOLD Responses in the rACC Cortex (Naltrexone vs Placebo)
Number analyzed (Participants) | 17
changes in BOLD signal | 1.23 (1.07)
Statistical Analysis 1: Comparison: fMRI BOLD Responses in the rACC Cortex (Naltrexone vs Placebo); Changes in BOLD fMRI signal from the Placebo vs. the Naltrexone session; Test type: Other — Mechanistic hypothesis: naltrexone will block contextual processing; p = 0.0002, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: [Approximately at day 1, 7]
Groups:
- Placebo: Placebo oral tablet: Placebo tablet that has no inherent power to produce an effect. In the inert pill condition, participants will receive an oral placebo tablet.
- Naltrexone: Naltrexone 50 Mg Oral Tablet: Naltrexone hydrochloride (ReVia®. Toronto, ON: Teva Canada Limited; 2015) (onset of action: ≥15 minutes; peak effect: ~1 hour; duration: ~24 hours).
Arm/Group | Placebo | Naltrexone
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 10/23 | 14/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | Naltrexone (N=24)
Nausea, gastrointestinal discomfort, vomiting. (Gastrointestinal disorders) | 3 (3) | 8 (8)
Fatigue (Nervous system disorders) | 6 (6) | 10 (10)
Dizziness/drowsiness (Nervous system disorders) | 4 (4) | 5 (5)
Shaking (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study does not have a healthy control condition, and therefore, results cannot be generalized beyond depression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT04322526/Prot_SAP_000.pdf